CLINICAL TRIAL: NCT00277316
Title: A Phase 2 Study of XL999 Administered Intravenously to Subjects With Metastatic Renal Cell Carcinoma
Brief Title: Study of XL999 in Patients With Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of XL999 was stopped due to cardiac toxicities in the subjects
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-201
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney cancer; Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — Treatment was administered on an outpatient basis. XL999 was administered at a dose of 2.4 mg/kg given as a 4 hour IV infusion.

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety, and tolerability of XL999 when given weekly to patients with metastatic clear cell renal cell carcinoma (RCC). XL999 is a small molecule inhibitor of multiple kinases including VEGFR, PDGFR, FGFR, FLT-3, and Src, which are involved in tumor cell growth, formation of new blood vessels (angiogenesis), and metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with histologically confirmed metastatic clear cell RCC
* Measurable disease according to Response Criteria for Solid Tumors (RECIST)
* No prior systemic cytotoxic chemotherapy
* Subjects who have received either no prior therapy for RCC, systemic immunotherapy only (such as interleukin-2 or interferon), or one agent targeting VEGF or a VEGFR (eg, bevacizumab, sorafenib, or sunitinib malate) may be enrolled
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months
* Adequate organ and marrow function
* No other malignancies within 5 years
* Signed informed consent

Exclusion Criteria:

* Radiation to ≥25% of bone marrow within 30 days of XL999 treatment
* Subjects who have received systemic anticancer therapy within 30 days of XL999 treatment
* Subjects who have not recovered to grade ≤1 or to within 10% of baseline from adverse events due to medications administered >30 days prior to study enrollment
* History of or known brain metastases, current spinal cord compression or carcinomatous meningitis
* Uncontrolled and/or intercurrent illness
* Pregnant or breastfeeding females
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Progression-free survival | Inclusion until disease progression
Duration of response | Inclusion until disease progression
Overall survival | Inclusion until 180-day Follow-up post last treatment or death
Pharmacokinetic (PK) and Pharmacodynamic (PD) parameters | Blood samples for PK/PD analysis will be obtained at the end of infusion for the first 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A. Bui, MD, Study Director — Exelixis
Locations (9):
- United States (9):
  - Department of Hematology/Oncology, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Integrated Community Oncology Network, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd, Joliet, Illinois
  - Division of Hematology/Oncology, Indiana University Cancer Center, Indianapolis, Indiana
  - The Cleveland Clinic Foundation Taussig Cancer Center, Cleveland, Ohio
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas